Effects of *Lentinula edodes* bar on lipid profile and antioxidant status in borderline high cholesterol individuals: a double blind randomized clinical trial

September 10th, 2019

## **Statistical Analysis**

Individuals data were stratified by gender, age, BMI, alcohol intake, physical activity and smoking. The differences between Shiitake and placebo groups were analyzed by the Chi-square test, Exact of Fisher test and Student's t-test.

Descriptions of all biochemical and oxidative stress parameters were expressed as mean  $\pm$  standard deviation. To investigate the differences in biochemical parameters between the groups, Analysis of Variance (ANOVA) with repeated measurements was applied. All results of biochemical parameters and oxidative stress were normalized to logarithmic scale. After normalization, statistical analysis was performed considering the differences among the intermediate and final times with the baseline. P < 0.05 was accepted as statistically significant. Data were analyzed using Stata® 14.2 software, College Station, Texas, USA.